CLINICAL TRIAL: NCT03664284
Title: Does the Disinfection of the Subcutaneous Tissue Reduce the Contamination of the Operative Field by P. Acnes During Primary Shoulder Surgery?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital du Valais (Other)
Responsible Party: Principal Investigator, Sina Grape, PD Dr Moor, Head of departement of orthopedic surgery, Principal investigator, Hôpital du Valais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-01269
Record Dates: First submitted 2018-09-07; First posted 2018-09-10 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Shoulder Surgery

STUDY DESIGN:
Intervention Model Description: The investigators will randomize 105 patient on two arms. The control group receiving no disinfection of the subcutaneous tissue (A) and intervention group, receiving disinfection of the subcutaneous tissue (B).
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator)
  Interventions: Procedure: subcutaneous disinfection
- control group (No Intervention)

INTERVENTIONS:
Procedure: subcutaneous disinfection — The investigators will randomize 105 patient on two arms. The control group receiving no disinfection of the subcutaneous tissue (A) and intervention group, receiving disinfection of the subcutaneous tissue (B).
  Arms: intervention group

SUMMARY:
Propionibacterium acnes is a pathogen frequently identified during postoperative infections of the shoulder. A recent study has shown that P. acnes is likely to be disseminated in the operative field from the subcutaneous layer by soft tissue manipulation by the surgeon and the instruments (Falconer 2016). This study seeks to evaluate the effectiveness of subcutaneous tissue disinfection on P. acnes contamination during primary shoulder surgery. The literature shows that approximately one-third of patients have a P. acnes-infected surgical drape during primary shoulder arthroplasty (Falconer 2016). The source of this contamination would be the subcutaneous tissue. The hypothesis is that a disinfection of the subcutaneous tissue would reduce the contamination of the operative field with the aim of reducing the infection rate after shoulder surgery.

DETAILED DESCRIPTION:
It is a randomized, single-center, open-label, category A clinical trial, a research project on people involved in the collection of biological material and the collection of health-related personal data with the existence of consent.

The investigators will study the effectiveness of Betadine subcutaneous tissue disinfection during primary shoulder surgery. They will randomize 105 patient on two arms. The control group receiving no disinfection of the subcutaneous tissue (A) and intervention group, receiving disinfection of the subcutaneous tissue (B). The investigators estimate that 4 years is enough to recruit the number of patients needed for this study.

All patients 18 years of age or older admitted to the Valais Hospital to receive primary shoulder surgery and who have signed the consent of the study will be eligible.

ELIGIBILITY:
Inclusion Criteria:

1. = or> 18 years
2. Supported at the Valais Hospital for primary surgery of the shoulder.
3. Have signed the consent

Exclusion Criteria:

1. <18 years old
2. History of shoulder surgery
3. History of infection of the shoulder
4. Antibiotherapy in the 2 weeks preceding the intervention
5. Infiltration of cortisone in the 6 months preceding the intervention
6. Iodinated contrast medium allergy or cefuroxime
7. Allergy to the povidone iodine complex or other contraindication to Betadine namely:

   Hypersensitivity to the active ingredient, iodine or povidone iodine complex, or to any of the excipients according to the composition.

   Hyperthyroidism and other overt thyroid diseases. Dermatitis herpetiformis of Duhring. Before and after radioactive iodine treatment (until the end of treatment)
8. Refusal of the terms of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
positive bacteriological sample | operation day
  To compare the positive bacteriological sample rate during open shoulder surgery with subcutaneous tissue disinfection compared to an identical procedure that does not include this step.

CONTACTS AND LOCATIONS:
Overall Officials: Beat K Moor, PD Dr, Principal Investigator — Hopital du Valais
Locations (1):
- Hopital du Valais, Martigny-Ville, Valais, Switzerland

REFERENCES:
- [Background] Falconer TM, Baba M, Kruse LM, Dorrestijn O, Donaldson MJ, Smith MM, Figtree MC, Hudson BJ, Cass B, Young AA. Contamination of the Surgical Field with Propionibacterium acnes in Primary Shoulder Arthroplasty. J Bone Joint Surg Am. 2016 Oct 19;98(20):1722-1728. doi: 10.2106/JBJS.15.01133. PMID 27869623